CLINICAL TRIAL: NCT02293525
Title: Investigational Plan for the Clinical Evaluation of the ReLeaf Analgesic Infusion Catheter & Wound Drain
Brief Title: Clinical Evaluation of the ReLeaf Analgesic Infusion Catheter & Wound Drain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were enrolled and the sponsor suspended support at this time
Sponsor: Vital 5, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLI-001-0201
Record Dates: First submitted 2014-10-27; First posted 2014-11-18 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Ropivacaine; Sodium Chloride; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Active Comparator): Continuous 0.2% Ropivacaine infusion until catheter removal (typically 36 hours)
  Interventions: Device: ReLeaf catheter; Drug: Ropivacaine; Drug: Morphine; Drug: Oxycodone
- Saline (Placebo Comparator): Continuous saline infusion until catheter removal (typically 36 hours)
  Interventions: Device: ReLeaf catheter; Drug: Saline; Drug: Morphine; Drug: Oxycodone

INTERVENTIONS:
Device: ReLeaf catheter — Continuous infusion rate 10ml/hr (5ml/side)
Drug: Ropivacaine
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Saline
  Arms: Saline
Drug: Morphine — Patient-controlled analgesia (PCA) at 1mg every 6 minutes with a 4 hour lock out after 30mg
Drug: Oxycodone — 10mg every 4-6 hours
  Other Names: Oxycontin, Roxicodone, Oxecta

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the ReLeaf infusion catheter & wound drain in patients following lumbar spinal fusion surgery. One half of the patients will receive continuous local analgesic fusion during the post-operative period while the other half will received continuous local saline.

DETAILED DESCRIPTION:
Posterior lumbar spinal fusion is commonly used in the management of a wide array of spinal disorders ranging from instability to degenerative disc disease. However, severe postoperative pain is a significant adverse outcome in patients who have undergone a lumbar spinal fusion procedure. This pain may delay mobilization and decrease compliance with physical, occupational, or pulmonary physiotherapy.

Pain symptoms may worsen with activity and ambulation due to reflex spasms of the paraspinal muscles elicited by pain from the wound. A local anesthetic agent administered immediately after surgery into the tissue surrounding the wound addresses the pain source for less than four hours. Therefore, it is reasonable to consider continuous local anesthetic infusion, which may limit local pain mediators for a longer duration.

Continuous local anesthetic infusion into the paraspinal musculature with the ReLeaf catheter has the potential to reduce pain, narcotic demand & usage, and accelerate the rate of recovery in lumbar spinal fusion patients.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Diagnosis of lumbar spine disease requiring an open, midline, instrumented posterolateral fusion with or without interbody support at one or two vertebral levels and laminectomy or laminotomy
* Physically and mentally willing to comply with the study requirements
* Signed the study informed consent

Exclusion Criteria:

* Lumbar spine disease requiring more than two levels of instrumentation
* Any previous operative lumbar procedure, except discectomy or hemi-laminotomy performed a minimum of 2 years prior to current study surgery
* Patients requiring iliac crest bone graft for the procedure
* Intra-operative durotomy
* Any duration of pre-operative morphine or morphine equivalent use exceeding 30 mg of morphine equivalents per day for longer than 3 months
* Physically or mentally compromised (i.e., being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease, presence of alcohol or substance abuse)
* Diagnosed with Severe Depression and on treatment
* Active infection at the operative level or a symptomatic infection
* Diagnosed systemic disease that would affect the subject's welfare or overall outcome of the research study (i.e. Paget's disease, renal osteodystrophy, Lupus etc)
* Is pregnant or breast feeding
* Has any active malignancy or spinal arthrodesis being performed for a tumor decompression
* Has a known allergy to local analgesics
* Pending litigation related to back pain or injury or Worker's Compensation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain (Mean VAS pain score at 24 hours post-procedure) | 24 hours
  Mean VAS pain score at 24 hours post-procedure

SECONDARY OUTCOMES:
Medication Use | 3 months
  Narcotic use from surgery through 3 months post-operative
Adverse Events | 3 months
  Occurrence of adverse events through 3 months post-operative

OTHER OUTCOMES:
Length of Hospital Stay | Discharge, on average 2 to 3 days
  Time from surgery to hospital discharge, on average 2 to 3 days
Incisional Pain | 3 months
  Pain at the site of the incision at 3 months post-operative
Incidence of nausea and vomiting | Discharge, on average 2 to 3 days
  Occurrence of nausea with or without vomiting and treatments from time of surgery through hospital discharge (which is 2-3 days on average)
Time of Foley Catheter Removal | Discharge, on average 2 to 3 days
  Time foley catheter was removed following surgery but no later than hospital discharge (which is 2-3 days on average)
Time to First Ambulate | Discharge, on average 2 to 3 days
  Time to walk following surgery but no later than hospital discharge (which is 2-3 days on average)

REFERENCES:
- [Background] Yukawa Y, Kato F, Ito K, Terashima T, Horie Y. A prospective randomized study of preemptive analgesia for postoperative pain in the patients undergoing posterior lumbar interbody fusion: continuous subcutaneous morphine, continuous epidural morphine, and diclofenac sodium. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2357-61. doi: 10.1097/01.brs.0000184377.31427.fa. PMID 16261108
- [Background] Gottschalk A, Freitag M, Tank S, Burmeister MA, Kreil S, Kothe R, Hansen-Algenstedt N, Weisner L, Staude HJ, Standl T. Quality of postoperative pain using an intraoperatively placed epidural catheter after major lumbar spinal surgery. Anesthesiology. 2004 Jul;101(1):175-80. doi: 10.1097/00000542-200407000-00027. PMID 15220788
- [Background] Bianconi M, Ferraro L, Ricci R, Zanoli G, Antonelli T, Giulia B, Guberti A, Massari L. The pharmacokinetics and efficacy of ropivacaine continuous wound instillation after spine fusion surgery. Anesth Analg. 2004 Jan;98(1):166-172. doi: 10.1213/01.ANE.0000093310.47375.44. PMID 14693613
- [Background] Elder JB, Hoh DJ, Wang MY. Postoperative continuous paravertebral anesthetic infusion for pain control in lumbar spinal fusion surgery. Spine (Phila Pa 1976). 2008 Jan 15;33(2):210-8. doi: 10.1097/BRS.0b013e318160447a. PMID 18197109